CLINICAL TRIAL: NCT05189769
Title: Reducing Racism and Discrimination in Schools: Comprehensive Prevention Services
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama, Tuscaloosa (Other)
Responsible Party: Principal Investigator, Sara McDaniel, PI; Professor, University of Alabama, Tuscaloosa
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 239047
Record Dates: First submitted 2021-11-30; First posted 2022-01-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Behavior, Child
Keywords: aggression; discipline
MeSH Terms: conditions — Child Behavior; Aggression

STUDY DESIGN:
Intervention Model Description: 2X2 randomized control trial across 2 districts
Who Masked: Participant
Masking Description: Design. This project will include a 5-year randomized control trial with four conditions: (a) PBIS and CP (serving as control), (b) SWPBIS+ and CP, (c) SWPBIS and CP+, and (d) SWPBIS+ and CP+.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CP/No REACT (Experimental): Traditional Coping Power for 7th graders, no school wide REACT training
  Interventions: Behavioral: CP no REACT
- CP/REACT (Experimental): Traditional Coping Power for 7th graders and school wide REACT training
  Interventions: Behavioral: CP and REACT
- CP+/No REACT (Experimental): New, adapted Coping Power for 7th graders intervention with no school wide REACT training
  Interventions: Behavioral: CP+/No REACT
- CP+/REACT (Experimental): New, adapted Coping Power for 7th graders, school wide REACT training
  Interventions: Behavioral: CP+ and REACT

INTERVENTIONS:
Behavioral: CP no REACT — Coping Power no REACT
  Arms: CP/No REACT
Behavioral: CP+/No REACT — CP+ and no REACT
  Arms: CP+/No REACT
Behavioral: CP and REACT — Coping Power traditional and REACT
  Arms: CP/REACT
Behavioral: CP+ and REACT — CP+ and REACT
  Arms: CP+/REACT

SUMMARY:
The primary purpose of this project is to test a comprehensive, two-part intervention with ReACT and a recently adapted, Coping Power+ Program. ReACT and PBIS are school-wide universal interventions. Coping Power and Coping Power+ are targeted preventive interventions designed to assist at-risk 7th grade students to improve their coping with interpersonal stressors during middle school. This project will evaluate the effects of the program on teacher, student and parent perceptions of school climate, student behavior, social-emotional competence, disciplinary infractions, and identity for 7th grade students in Coping Power or Coping Power+

DETAILED DESCRIPTION:
Project Rationale Data from public Middle Schools indicate increasing rates of unsafe, disruptive, and event violent behaviors across the US. These incidents may also include peer victimization. Racially and ethnically minoritized youth are disproportionately affected by these incidents and occurrences of racial bias in school. The purpose of the Comprehensive Prevention Strategies (CPS) intervention is to preventatively promote youth safety and belonging across individual, school, and community settings by intervening at multiple entry points. The primary components include: (1) an adapted version of Coping Power and (2) extended PBIS strategies called "ReACT" (Racial equity through Assessing data for vulnerable decision points, culturally responsive behavior strategies, and Teaching about implicit bias and how to neutralize it) is for teachers. This project leverages the evidence-based Coping Power student and parent interventions and Positive Behavioral Interventions and Supports (PBIS) approaches to include much-needed adaptations to address this critical issue. This project has the potential for important public health outcomes: (a) reducing youth violence, (b) improving school climate and (c) improving teacher practices regarding discipline, disproportionate discipline, and bias in public schools.

Project Aims The primary purpose of this project is to test a comprehensive, two-part intervention with ReACT and a recently adapted, Coping Power+ Program. ReACT and PBIS are school-wide universal interventions. Coping Power and Coping Power+ are targeted preventive interventions designed to assist at-risk 7th grade students to improve their coping with interpersonal stressors during middle school. This project will evaluate the effects of the program on teacher, student and parent perceptions of school climate, student behavior, social-emotional competence, disciplinary infractions, and identity for 7th grade students in Coping Power or Coping Power+

Funding This project is funded by a 5-year grant awarded by the National Institute of Minority Health and Health Disparities.

Sample of Schools A total of 18 middle schools have been recruited for involvement in this project: 11 in Huntsville City Schools and 7 in Jefferson County Public Schools.

Student Participation and Data Collection Students who are identified by teachers and/or school staff as potentially benefiting from Coping Power on the 6-item universal screener completed by 6th grade teachers each project year in the spring, will be contacted by school staff to request active parental consent for participation.

Benefits to Participating Schools To implement the Coping Power and Coping Power+ Programs, clinicians will be hired by the grant and will be co-trained with one or more school-based staff members (e.g., school counselor, school psychologist). In appreciation of staff time devoted to leading the Coping Power groups, the grant will provide a $25 per session donation to the school ($625 per year).

This project will increase the school's capacity to implement an evidence-based Tier 3 prevention program to support students and their families.

Timeline This 5-year project began in 2019 with the development of CP+ adaptations and ReACT strategies for middle school. Study activities were halted in 2020 due to the pandemic. In August of 2021 researchers will continue with ReACT educator training (on full day), then send parental permission forms for Coping Power participation. Coping Power groups will start in September and run weekly for the rest of the year. ReACT training will be followed by monthly one-hour strategy sessions for the remainder of the school year. While ReACT training will be complete, another cohort of 7th grade students will enter Coping Power (screened in each spring) in September 2022 and September 2023. Each year approximately 17 students from each middle school will participate in Coping Power groups.

Expected Outcome Researchers proposed that adapted, culturally responsive Coping Power will be more effective than traditional Coping Power in promoting prosocial behavior for 7th grade participants.

ReACT Teacher Training

ReACT (Racial equity through Assessing data for vulnerable decision points, Culturally responsive behavior strategies, and Teaching about implicit bias and how to neutralize it) is a universal professional development intervention for all school staff to leverage the PBIS framework for increasing racial equity in school discipline (McIntosh, Barnes, et al., 2014). The intervention includes whole-school professional development sessions delivered throughout the year that focus on understanding discipline decision making and the effects of bias, a root cause analysis of discipline data, and creation of a tailored intervention plan with strategies selected to address these root causes.

Middle School Coping Power Child and Parent Program The Coping Power Program is a rigorously tested, multi-component school-based intervention for children and their parents (Lochman & Wells, 1996), that addresses issues related to aggression and problem behavior. Efficacy and effectiveness studies conducted in multiple schools in Alabama and throughout the United States over the past two decades have found Coping Power to reduce students' levels of externalizing and internalizing behaviors, and substance use, and to enhance students' language artss grades through long-term follow-up periods, in comparison to randomized control and comparison students. families in need of specialized services.

The Coping Power student component is offered to groups of six students at the school and features 25 weekly group sessions, each lasting about 45 minutes. The program includes 12 parenting sessions during which parents meet in groups of 10-12 with two co-leaders.

Aim 1. To determine the extent to which SWPBIS+ training is more effective than SWPBIS alone as a Tier 1, in reducing disproportionate disciplinary practices, and if differences are moderated by student and teacher race.

Aim 2. To determine the extent to which CP+ is more effective than CP as a targeted intervention in reducing interracial and intraracial aggression and if differences are moderated by student race.

Aim 3. To determine the extent to which the effects of CP+ relative to CP differ depending on the Tier 1 context (SWPBIS+ vs. SWPBIS) and whether those effects are moderated by student race.

In addition, poverty will be included as potential covariates in the model at both the individual (student free/reduced price lunch status) and school (percentage of students receiving free/reduced price lunch) levels.

ELIGIBILITY:
Inclusion Criteria:

* 7th grader
* screened on NIDA screener as in the highest 25 percentile on risk in target school

Exclusion Criteria:

* None

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1093 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
National Institute on Drug Abuse Quick Screener: Teacher Report of Reactive and Proactive Behaviors. | Pre-intervention
  his 6-item screener will be completed on all students in participating classrooms. Higher scores indicate more risk to determine the top 25% of the scoring students who will be considered participants in the CP and CP+ groups. T
Behavior Assessment Scale for Children (BASC)-Third Edition Teacher Report Scale Child Form (BASC-3). | Pre-intervention
  The BASC-3 Teacher Rating Scale has 139 items and takes approximately 15 minutes to complete. Higher scores indicate more risk
School Climate | Pre-intervention and immediately after intervention concludes
  he Georgia School Climate Survey (GSCS) is a computerized school climate rating scale that was developed as part of the Georgia School Climate Survey Suite (Georgia Department of Education, La Salle, Meyers, 2014).

SECONDARY OUTCOMES:
Discipline Incidents. | immediately after intervention concludes
  An office discipline referral (ODR) represents an incident (i.e., major infraction) in which a student was observed by a staff member violating a school rule or social norm and then provided a consequence by an administrator who made a permanent record of the event

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Jefferson County Public Schools, Birmingham, Alabama
  - Huntsville City Schools, Huntsville, Alabama

IPD SHARING:
Plan to Share IPD: No
No plan at this time